CLINICAL TRIAL: NCT02548195
Title: Oxaliplatin Plus Gemcitabine Versus Capecitabine Alone as Adjuvant Treatment in the Prevention of Recurrence of Intrahepatic Cholangiocarcinoma
Brief Title: Oxaliplatin+Gemcitabine vs Capecitabine as Adjuvant Therapy for Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Vice Director of the Department of Liver Surgery, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gemoxicc
Record Dates: First submitted 2015-08-07; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Cholangiocarcinoma
Keywords: GEMOX; intrahepatic cholangiocarcinoma; adjuvant therapy; oxaliplatin; gemcitabine; capecitabine; curative surgery
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Oxaliplatin; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GEMOX (Experimental): oxaliplatin and gemcitabine (GEMOX regimen): day 1: oxaliplatin 85 mg/m2, gemcitabine 1000 mg/m2; day 8: gemcitabine 1000 mg/m2; every three weeks for 6-8 cycles in total.
  Interventions: Drug: oxaliplatin and gemcitabine
- Capecitabine (Active Comparator): capecitabine 1250 mg/m2, twice daily for two weeks plus one week rest for 8 cycles in total.
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: oxaliplatin and gemcitabine — oxaliplatin and gemcitabine (GEMOX regimen): day 1: oxaliplatin 85 mg/m2, gemcitabine 1000 mg/m2; day 8: gemcitabine 1000 mg/m2 every three weeks for 6-8 cycles in total.
  Other Names: oxaliplatin; gemcitabine
  Arms: GEMOX
Drug: capecitabine — capecitabine 1250 mg/m2, twice daily for two weeks plus one week rest for 8 cycles in total.
  Other Names: Xeloda
  Arms: Capecitabine

SUMMARY:
To evaluate of adjuvant therapy using oxaliplatin and gemcitabine (GEMOX regimen) versus capecitabine alone chemotherapy in patients who underwent curative surgery for intrahepatic cholangiocarcinoma (ICC) -- a randomized control study.

DETAILED DESCRIPTION:
chemotherapy: GEMOX vs capecitabine alone; adjuvant settings; primary endpoint: recurrence-free survival (RFS); second endpoint: overall survival after surgery (OS).

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS≤1;
* pathologically confirmed adenocarcinoma of bile duct;
* R1 resection or R0 resection with these risk factors: lymph node metastasis, lymphatic vessel or blood vessel invasion, multiple tumors, tumor size >5 cm, preoperative CA199>200 U/mL.
* postoperative liver function Child Pugh Class A, leukocyte count>1.5*10^9/L, platelet count>100*10^9/L, serum alanine aminotransferase <1.5*ULN
* no tumor recurrence or metastasis on baseline examination
* no history of radiotherapy or intervention therapy

Exclusion Criteria:

* hepatocellular carcinoma, mixed carcinoma of ICC and HCC, or hilar cholangiocarcinoma
* distant metastasis
* prothrombin time >14s
* severe cardiopulmonary dysfunction
* severe renal dysfunction
* bone marrow suppression before the initiation of therapy
* allergic to fluorouracil, gemcitabine, or platinum
* gemcitabine was used in combination with radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | from the date of surgery to the date of tumor recurrence up to 36 months after surgery

SECONDARY OUTCOMES:
Overall survival | from the date of surgery to the date of death up to 36 months after surgery

OTHER OUTCOMES:
Number of participants with adverse events and severe adverse events | from the date of first dosage to safety follow-up visit (30 days after the last dosage)
  All toxicities will be graded by CTCAE v4

CONTACTS AND LOCATIONS:
Overall Officials: Jinpei Huang, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Result] Cho SY, Park SJ, Kim SH, Han SS, Kim YK, Lee KW, Lee SA, Hong EK, Lee WJ, Woo SM. Survival analysis of intrahepatic cholangiocarcinoma after resection. Ann Surg Oncol. 2010 Jul;17(7):1823-30. doi: 10.1245/s10434-010-0938-y. Epub 2010 Feb 18. PMID 20165987
- [Result] Schmoll HJ, Twelves C, Sun W, O'Connell MJ, Cartwright T, McKenna E, Saif M, Lee S, Yothers G, Haller D. Effect of adjuvant capecitabine or fluorouracil, with or without oxaliplatin, on survival outcomes in stage III colon cancer and the effect of oxaliplatin on post-relapse survival: a pooled analysis of individual patient data from four randomised controlled trials. Lancet Oncol. 2014 Dec;15(13):1481-1492. doi: 10.1016/S1470-2045(14)70486-3. Epub 2014 Nov 12. PMID 25456367
- [Result] Patt YZ, Jones DV Jr, Hoque A, Lozano R, Markowitz A, Raijman I, Lynch P, Charnsangavej C. Phase II trial of intravenous flourouracil and subcutaneous interferon alfa-2b for biliary tract cancer. J Clin Oncol. 1996 Aug;14(8):2311-5. doi: 10.1200/JCO.1996.14.8.2311. PMID 8708722
- [Result] Ducreux M, Van Cutsem E, Van Laethem JL, Gress TM, Jeziorski K, Rougier P, Wagener T, Anak O, Baron B, Nordlinger B; EORTC Gastro Intestinal Tract Cancer Group. A randomised phase II trial of weekly high-dose 5-fluorouracil with and without folinic acid and cisplatin in patients with advanced biliary tract carcinoma: results of the 40955 EORTC trial. Eur J Cancer. 2005 Feb;41(3):398-403. doi: 10.1016/j.ejca.2004.10.026. PMID 15691639
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404